CLINICAL TRIAL: NCT06060561
Title: Genetic Testing to Improve Management of Patients Undergoing Breast Biopsy
Status: Suspended | Type: Observational
Why Stopped: on hold for analysis
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 22-011193; NCI-2023-06044 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 22-011193 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2023-09-22; First posted 2023-09-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational: Patients undergo saliva sample collection and complete questionnaires on study. Patients' medical records are reviewed.
  Interventions: Other: Non-Interventional Study

INTERVENTIONS:
Other: Non-Interventional Study — Non-interventional study

SUMMARY:
This study evaluates genetic testing to improve risk assessment and advance efforts to develop precision management for breast cancer by studying saliva samples for genotyping and evaluate associations with pathologic diagnoses and detailed pathologic and radiologic features.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To collect saliva from 500 consenting women undergoing a clinically indicated breast biopsy, perform genotyping, and then assess the associations of polygenic risk score (PRS) (and related single nucleotide polymorphisms [SNPs]) to final diagnosis of ductal carcinoma in situ (DCIS), invasive breast cancer or benign breast disease (BBD); BBD severity; specific BBD lesions; and features of background benign lobules from which these lesions arise.

II. To relate PRS (and related SNPs) to radiologic features, including breast density and sentinel lesions, such as masses, densities, calcifications, and asymmetries.

III. To relate PRS (and related SNPs) to molecular markers in pathologic lesions and background tissues, including associations with breast cancer (BC) molecular subtypes (e.g., luminal, triple-negative (basal) and human epidermal growth factor receptor 2 [HER2] overexpressing) and biomarkers in BBD and lobules.

OUTLINE: This is an observational study.

Patients undergo saliva sample collection and complete questionnaires on study. Patients' medical records are reviewed.

ELIGIBILITY:
Inclusion Criteria:

* * Women over the age of 18 years

  * Able to provide informed consent
  * Referred for a radiologically guided breast biopsy

Exclusion Criteria:

* * Men

  * Women under the age of 18 years
  * Unable to provide informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women referred for a radiologically guided breast biopsy.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-05-30 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of subjects consented per month | Baseline; Up to study completion (approximately 5 years)
  Will be assessed by the percentage of eligible patients consented.
Deoxyribonucleic acid (DNA) quantity | Up to study completion (approximately 5 years)
  Will analyze DNA from saliva sample to assess quantity for a validated polygenic risk score (PRS) for breast cancer.
Deoxyribonucleic acid (DNA) quality | Up to study completion (approximately 5 years)
  Will analyze DNA from saliva sample to assess quality for a validated PRS for breast cancer.
Ability to perform genotyping using collected sample | Up to study completion (approximately 5 years)
  Will perform genotyping on collected saliva sample using the Infinium Global Diversity Array test to generate a validated polygenic risk score (PRS) for breast cancer. Test results will be reviewed to assess whether the saliva sample contains enough (quantity) viable (quality) deoxyribonucleic acid (DNA) to provide accurate genotype results.
Success in estimation of polygenic risk score (PRS) | Up to study completion (approximately 5 years)
  Medical records will be reviewed and compared with study findings to determine success of PRS estimation.

CONTACTS AND LOCATIONS:
Overall Officials: Mark E. Sherman, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials